CLINICAL TRIAL: NCT06035770
Title: The Effectiveness of Ensa - Mental Health First Aid Training on Knowledge and Mental Health of Undergraduate Students in Switzerland: a Randomised Control Trial.
Brief Title: The Effectiveness of Mental Health First Aid Intervention Among Undergraduate Students in Switzerland
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut et Haute Ecole de la Santé la Source (Other)
Collaborators: HEIG-VD- Haute Ecole d'Ingénierie et de Gestion du Canton de Vaud (Unknown)
Responsible Party: Principal Investigator, Meichun Mohler-Kuo, Sc.D, Sc.D. Professeur Ordinaire HES-SO, Institut et Haute Ecole de la Santé la Source
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2019-01296
Record Dates: First submitted 2023-06-23; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Preventative Medicine
Keywords: mental health first aid;; undergraduate students;; RCT; intervention; education program

STUDY DESIGN:
Intervention Model Description: Randomized Control trial with educational intervention
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mental Health First Aid training program (Experimental): The intervention is a 12-hour face-to-face training course given in small groups. It was delivered as four 3-hour sessions over 4 consecutive weeks.
  Interventions: Other: Mental Health First Aid (educational training program)
- control group (No Intervention): The control group received no intervention during the intervention period. However, they will participate in surveys at three time points (before the intervention, 3 months after the intervention and one year after the intervention). Once their final assessment is completed, controls will be offered the opportunity to take the MHFA training course, if they wish.

INTERVENTIONS:
Other: Mental Health First Aid (educational training program) — The MHFA program is a 12-hour face-to-face training program delivered in four sessions of three hours each across four consecutive weeks by two accredited MHFA instructors. The class was administered in small groups with a maximum of 10-15 students.The program included didactic lectures and "role playing" to teach students how to recognize and react to the signs and symptoms of mental health illness. Participants enrolled in the intervention group received an accompanying manual with content that covered helping people in mental health crises and/or the early stages of mental health problems.
  The mental health problems addressed during the training session included depressive symptoms, anxiety, psychotic disorders, and substance use disorders. The mental health crisis situations included suicidal thoughts/attempts and behaviors, acute stress reactions,panic attacks, and acute psychotic behaviors.
  Arms: Mental Health First Aid training program

SUMMARY:
Mental Health First Aid (MHFA) is an educational training program which has been proven effective at increasing knowledge, improving attitudes and reducing the stigma of mental illness among individuals/the general population. Although MHFA has proven effective world-wide, no study has examined the effectiveness of MHFA in Switzerland and very few studies have examined the long-term effects of MHFA and how they might be influenced by cultural differences. This study is a randomized control trial (RCT) that examines the effectiveness of a 12-hour MHFA training program that aims to improve undergraduate students' knowledge of, behaviours towards mental illness and to reduce stigmatization towards mental illness. All participants were 2nd-year students and they were randomly assigned either to an intervention group that would receive the MHFA training course or to a control group without any intervention during the study period. However, the control group had the option to receive the MHFA course after the 12 months of study follow-up was completed. Both groups were assessed at three time points: T0: Baseline survey from mid-September to October 2019, completed by both groups.

Intervention: MHFA training program from October 2019-December 2019. T1: Post-intervention with first follow-up survey three months after the MHFA training intervention completed by both groups (from March to May 2020). T2: Follow-up 12 months after the MHFA/ensa training intervention in December 2020 and completed by both groups.

ELIGIBILITY:
Inclusion Criteria:

* 2nd year undergraduate students from universities of applied science in Lausanne and Yverdon-les-Bains.
* ≥18 years old.

Exclusion Criteria:

* Working and part-time students.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2019-09-20 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Level of knowledge-(changes were assessed at 3 and 12 months) | 3 months; 12 months
  to measure participants' ability to identify a mental health problem and answer questions based on the content of the MHFA course. Changes of knowledge level before and after the MHFA intervention are also assessed.
Level of attitudes pertaining to mental illness (changes were assessed at 3 and 12 months) | 3 months; 12 months
  to measure changes of participants' level of stigmatization and social distance toward mental illness. Changes of before and after the intervention are also assessed.
behaviors toward mental illness (changes are assessed at 3 and 12 months)) | 3 months; 12 months
  to measure participants' confidence and intention to provide help and the changes before and after the MHFA are also assessed.

SECONDARY OUTCOMES:
mental health-quality of life (changes were assessed assessed at 3 and 12 months) | 3 months; 12 months
  Quality of life using Short-Form Health Survey (SF-12) and change of quality of life were assessed.
mental health-depression (changes were assessed at 3 and 12 months) | 3 months; 12 months
  Depression symptoms ( using Patient Health Questionnaire (Brief PHQ-9) and change of depression symptoms were assessed.
change of mental health-anxiety | 3 months; 12 months
  Anxiety symptom (using Generalized Anxiety Disorder 7) and changes of anxiety symptoms were assessed.
change of mental health-ADHD symptoms | 3 months; 12 months
  ADHD symptoms were assessed using 'ADHD Self-Report Scale (ASRS)' Screener and the change of ADHD symptoms was also assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Meichun Mohler-Kuo, Sc.D., Principal Investigator — La Source, School of Nursing Sciences, HES-SO
Locations (1):
- La Source, School of Nursing Sciences, HES-SO University of Applied Sciences Western Switzerland., Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dzemaili S, Pasquier J, Oulevey Bachmann A, Mohler-Kuo M. The Effectiveness of Mental Health First Aid Training among Undergraduate Students in Switzerland: A Randomized Control Trial. Int J Environ Res Public Health. 2023 Jan 11;20(2):1303. doi: 10.3390/ijerph20021303. PMID 36674060